CLINICAL TRIAL: NCT01699204
Title: Effects of Diesel Exhaust on Airways
Brief Title: Diesel Exhaust and Mechanism of Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Christopher Carlsten, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: H08-02288
Record Dates: First submitted 2012-10-01; First posted 2012-10-03 (Estimated); Last update posted 2017-09-29 (Actual); Status verified 2017-09

CONDITIONS: Asthma
Keywords: Air pollution; Diesel exhaust; Airway responsiveness; Asthma; Anti-oxidant
MeSH Terms: conditions — Asthma | interventions — Acetylcysteine; Vehicle Emissions

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Filtered air with placebo (Placebo Comparator): Exposure for 2 hours to filtered air and placebo tablets 3 times daily for 6 days
  Interventions: Other: Filtered air
- Diesel exhaust with placebo (Active Comparator): Exposure for 2 hours to diesel exhaust and placebo tablets 3 times daily for 6 days
  Interventions: Other: Diesel exhaust
- Diesel exhaust with N-acetylcysteine (Experimental): Exposure for 2 hours to diesel exhaust and N-acetylcysteine tablets (600 mg) 3 times daily for 6 days
  Interventions: Dietary Supplement: N-acetylcysteine; Other: Diesel exhaust

INTERVENTIONS:
Dietary Supplement: N-acetylcysteine — N-acetylcysteine 600mg taken orally 3 times daily for 6 days prior to exposure to diesel exhaust for 2 hours. The last supplement was taken the morning of the exposure
  Arms: Diesel exhaust with N-acetylcysteine
Other: Diesel exhaust — A placebo tablet taken 3 times daily for 6 days prior to exposure to diesel exhaust for 2 hours. The last supplement was taken the morning of the exposure
  Arms: Diesel exhaust with N-acetylcysteine; Diesel exhaust with placebo
Other: Filtered air — A placebo tablet taken 3 times daily for 6 days prior to exposure to filtered air for 2 hours. The last supplement was taken the morning of the exposure
  Arms: Filtered air with placebo

SUMMARY:
This experiment is designed to test the hypothesis that oxidative stress is responsible for changes in airway responsiveness in humans exposed to diesel exhaust.

DETAILED DESCRIPTION:
The specific aim is to test the hypothesis that diesel exhaust (DE) increases airway reactivity via oxidative stress, particularly in asthmatics. To test this hypothesis, we use a crossover in vivo experimental model in mild asthmatics and normal controls using a state-of-the-art diesel exhaust exposure facility.

Participants took N-acetylcysteine (600 mg) or placebo capsules three times daily for six days. On the final morning of supplementation, participants were exposed for 2 hours to either filtered air or diesel exhaust (300 µg·m-3 of particulate matter smaller than 2.5 microns). Twenty-six non-smokers between 19-49 years were studied under three experimental conditions (filtered air with placebo, diesel exhaust with placebo and diesel exhaust with N-acetylcysteine) using randomized, double-blind, crossover design, with a two week minimum washout between conditions. Methacholine challenge was performed pre-exposure (to determine baseline airway responsiveness) and post-exposure (to determine the effect of exposure).

ELIGIBILITY:
Inclusion Criteria:

* Between 19-49 years, non smokers, asthmatics, healthy controls

Exclusion Criteria:

* Smokers, pregnant or co-existing medical condition for which diesel exhaust would confer significant risk (i.e. coronary artery disease)

Ages: 19 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2007-09; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Human airway reactivity | 50 hours
  Establish that oxidative stress is responsible for changes in human airway reactivity induced by DE (300 µg/m3 inhaled for two hours).

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Carlsten, MD MPH, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia, Vancouver, British Columbia, Canada

REFERENCES:
- [Background] Braman SS. The global burden of asthma. Chest. 2006 Jul;130(1 Suppl):4S-12S. doi: 10.1378/chest.130.1_suppl.4S. PMID 16840363
- [Background] Atkinson RW, Anderson HR, Sunyer J, Ayres J, Baccini M, Vonk JM, Boumghar A, Forastiere F, Forsberg B, Touloumi G, Schwartz J, Katsouyanni K. Acute effects of particulate air pollution on respiratory admissions: results from APHEA 2 project. Air Pollution and Health: a European Approach. Am J Respir Crit Care Med. 2001 Nov 15;164(10 Pt 1):1860-6. doi: 10.1164/ajrccm.164.10.2010138. PMID 11734437
- [Background] Janssen NA, Brunekreef B, van Vliet P, Aarts F, Meliefste K, Harssema H, Fischer P. The relationship between air pollution from heavy traffic and allergic sensitization, bronchial hyperresponsiveness, and respiratory symptoms in Dutch schoolchildren. Environ Health Perspect. 2003 Sep;111(12):1512-8. doi: 10.1289/ehp.6243. PMID 12948892
- [Background] Mudway IS, Stenfors N, Duggan ST, Roxborough H, Zielinski H, Marklund SL, Blomberg A, Frew AJ, Sandstrom T, Kelly FJ. An in vitro and in vivo investigation of the effects of diesel exhaust on human airway lining fluid antioxidants. Arch Biochem Biophys. 2004 Mar 1;423(1):200-12. doi: 10.1016/j.abb.2003.12.018. PMID 14871482
- [Background] Rudell B, Ledin MC, Hammarstrom U, Stjernberg N, Lundback B, Sandstrom T. Effects on symptoms and lung function in humans experimentally exposed to diesel exhaust. Occup Environ Med. 1996 Oct;53(10):658-62. doi: 10.1136/oem.53.10.658. PMID 8943829
- [Background] Stenfors N, Nordenhall C, Salvi SS, Mudway I, Soderberg M, Blomberg A, Helleday R, Levin JO, Holgate ST, Kelly FJ, Frew AJ, Sandstrom T. Different airway inflammatory responses in asthmatic and healthy humans exposed to diesel. Eur Respir J. 2004 Jan;23(1):82-6. doi: 10.1183/09031936.03.00004603. PMID 14738236
- [Background] Hashimoto S, Gon Y, Takeshita I, Matsumoto K, Jibiki I, Takizawa H, Kudoh S, Horie T. Diesel exhaust particles activate p38 MAP kinase to produce interleukin 8 and RANTES by human bronchial epithelial cells and N-acetylcysteine attenuates p38 MAP kinase activation. Am J Respir Crit Care Med. 2000 Jan;161(1):280-5. doi: 10.1164/ajrccm.161.1.9904110. PMID 10619832
- [Background] McCreanor J, Cullinan P, Nieuwenhuijsen MJ, Stewart-Evans J, Malliarou E, Jarup L, Harrington R, Svartengren M, Han IK, Ohman-Strickland P, Chung KF, Zhang J. Respiratory effects of exposure to diesel traffic in persons with asthma. N Engl J Med. 2007 Dec 6;357(23):2348-58. doi: 10.1056/NEJMoa071535. PMID 18057337